CLINICAL TRIAL: NCT03522480
Title: The Effectiveness of the Jamboxx Respiratory Therapy Device in Treatment of Patients With Decreased Respiratory Function. Study 2: Children With Cystic Fibrosis for Long Term Evaluation
Brief Title: The Effectiveness of the Jamboxx Respiratory Therapy Device: Study 2
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Change of Research Objectives for Grant Funded Study
Sponsor: My Music Machines Inc. (Industry)
Collaborators: Albany Medical College (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Jamboxx RT Device Study 2; 4R42HL132735-02 (NIH)
Record Dates: First submitted 2018-04-26; First posted 2018-05-11 (Actual); Last update posted 2020-09-02 (Actual); Status verified 2019-01

CONDITIONS: Cystic Fibrosis in Children
Keywords: cystic fibrosis; autogenic drainage; respiratory therapy; videogaming therapy
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of two study groups: A or B. Participants assigned to study group A will be taught by a respiratory therapist how to perform the autogenic drainage technique in week 0, and will be asked to perform the technique regularly on their own for secretion clearance for the first 8 weeks of the study. Beginning in week 8, they will be taught to use autogenic draining technique guided by a videogame through the Jamboxx respiratory therapy device and will be advised to perform the technique regularly using the game for guidance through week 16 Participants in group B will be taught to perform the autogenic draining technique using the Jamboxx respiratory therapy guided by a videogame in week 0, and will be instructed to perform the technique regularly for the next 16 weeks using the game for guidance
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Group A: Education & Gaming (Other): Children will participate in 1 initial training session where they will be taught by a RT to use autogenic drainage (AD). Patients will be sent home & prescribed to practice the technique 15 minutes 3 times / week. At week 8 +/- 1 week patients will return and will be tested by a software program designed to evaluate their ability to perform the AD sequence (percent accuracy). At the 8 week visit, the Jamboxx gaming device will be introduced, which will contain a game to guide them through the proper sequence of breathing for the AD technique. Patients will be sent home with a Jamboxx device and requested to do 15 minutes of AD training 3 times / week. Patients will return at week 16 and again will be tested via software program for ability to perform the AD technique.
  Interventions: Device: Jamboxx Respiratory Therapy Device; Other: Autogenic Draining Training
- Group B: Gaming Only (Experimental): Children will participate in an initial training session at Albany Med where they will be taught by a RT to use the Jamboxx respiratory therapy device to guide them through autogenic drainage (AD): a series of controlled breathing exercises that mobilizes mucous without inducing wheezing in patients with reactive airways. Patients will be sent home and prescribed to use the Jamboxx respiratory therapy device 15 minutes three times per week. At week 8 and week 16 +/- 1 week patients will return and will be tested by a software program designed to evaluate their ability to perform AD sequence (percent accuracy).
  Interventions: Device: Jamboxx Respiratory Therapy Device

INTERVENTIONS:
Device: Jamboxx Respiratory Therapy Device — The Jamboxx Respiratory Therapy Device is a novel device that uses interactive gaming to encourage patient compliance with their prescribed respiratory therapy routines. The device consists of a computer game controller with mouthpiece, and breath flow sensor that connects to a tablet. With the Jamboxx respiratory therapy device, users can choose from a suite of breath controlled respiratory therapy games to guide them through their routines while receiving real-time feedback, and long-term progress tracking.
Other: Autogenic Draining Training — A respiratory therapist will teach children how to conduct the autogenic draining technique (a series of exhalations and inhalations) by demonstrating the technique to them, and having them practice in their office. Children will also receive an informational packet and short video about the technique for reference
  Arms: Group A: Education & Gaming

SUMMARY:
The Effectiveness of the Jamboxx Respiratory Therapy Device in Treatment of Patients with Decreased Respiratory Function is a proposal for investigation of the application of gaming to improving respiratory health. The Jamboxx device combines gaming with traditional incentive spirometry to provide users with a fun experience to keep them engaged in their respiratory therapy routine. The device allows users to play a series of mini-games that walk them through their routines. The Jamboxx also records airflow and lung parameters with an external mouthpiece attachment to provide users with real time feedback, and helps to assess increases or decreases in relative lung function over time. The Jamboxx has the potential to significantly impact the field of respiratory therapy by being one of the first gaming devices for patient therapy, and the first respiratory therapy gaming device that is accessible to users with limited mobility. Jamboxx provides a fun and engaging, low cost alternative to the traditional therapy techniques used and aims to improve patient compliance.

This study addresses the ongoing challenge of clearing the burden of bronchial secretions resulting from cystic fibrosis. These patients are dependent upon mechanical devices to help clear secretions. A device autonomous means for clearing secretions is well defined in the literature (autogenic drainage) but is difficult to learn. This study proposes to teach cystic fibrosis patients to master autogenic drainage, and seeks to determine at what age it can be taught. As it would be expected that gaming could easily teach adults this procedure, the study will include children for whom learning autogenic drainage based upon conceptualization would be expected to be very difficult.

DETAILED DESCRIPTION:
Testing Plan: Children will be randomized into one of two groups via a random number generation software program

Group A (education & gaming): Children will participate in 1 initial training session at Albany Med where they will be taught by a respiratory therapist (RT) to use autogenic drainage: a series of controlled breathing exercises that mobilizes mucous without inducing wheezing in patients with reactive airways. Patients will be sent home and prescribed to practice the autogenic draining technique 15 minutes three times per week. At week 8 +/- 1 week patients will return for study visits and will be tested by a software program designed to evaluate their ability to perform autogenic drainage sequence (percent accuracy). This will be done through a software program installed on the device that uses a series of calibration breaths to fit a curve that models the individual patient's idealized autogenic drainage sequence, then maps their actual performance to this curve and calculates a percent accuracy. At the 8 week visit, the Jamboxx gaming device will be introduced through a training session with a RT, which will contain a game to guide them through the proper sequence of breathing for the autogenic draining technique. Patients will be sent home with a Jamboxx device and requested to do 15 minutes of autogenic drainage training three times a week. Patients will return for a research visits at week 16 and again will be tested via software program for ability to perform the autogenic drainage technique.

Group B (gaming only): Children will participate in an initial training session at Albany Med where they will be taught by a RT to use Jamboxx respiratory thearpy device to guide them through autogenic drainage: a series of controlled breathing exercises that mobilizes mucous without inducing wheezing in patients with reactive airways. Patients will be sent home and prescribed to use the Jamboxx respiratory therapy device 15 minutes three times per week. At week 8 and week 16 +/- 1 week patients will return for study visits and will be tested by a software program designed to evaluate their ability to perform autogenic drainage sequence (percent accuracy). This will be done through a software program installed on the device that uses a series of calibration breaths to fit a curve that models the individual patient's idealized autogenic drainage sequence, then maps their actual performance to this curve and calculates a percent accuracy.

This protocol does not replace prescribed chest physiotherapy. There is no alteration of the standard of care beyond 15 minutes of autogenic drainage three times per week. Demographic data (age, gender, ethnicity) will be collected. Medical records will be evaluated for relevant health history, medication use, and hospitalizations including dates.

ELIGIBILITY:
Inclusion Criteria:

* Children with CF requiring chest physiotherapy ages 5-17

Exclusion Criteria:

* Children with lung function of <25% FEV, hypercapnia, or requiring supplemental oxygen will be excluded.

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2019-01-30 (Actual); Primary Completion 2019-08-31 (Estimated); Study Completion 2019-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in accuracy with the autogenic draining technique | Weeks 0, 8, 16
  A software program has been developed by the study team to evaluate ability to perform autogenic drainage sequence (percent accuracy). This program will be installed on the Jamboxx Respiratory Therapy device (without the associated games), and uses a series of calibration breaths to fit a curve that models the individual patient's idealized autogenic drainage sequence, then maps their actual performance to this curve and calculates a change in percent accuracy from the baseline value to the end of the 16 week study.

SECONDARY OUTCOMES:
Cystic Fibrosis Questionnaire- Revised | Weeks 0, 16
  A study developed by the Cystic Fibrosis Foundation to evaluate respiratory function and overall health and wellbeing for children living with CF
Clinically relevant events & exacerbations | Weeks 0, 8, 16
  e.g. patient being sent for a chest x-ray, being ordered chest physiotherapy, prescribed to new systemic antibiotics, hospital admission

CONTACTS AND LOCATIONS:
Overall Officials: Marilyn Fisher, MD, Study Chair — Albany Medical Center IRB
Locations (1):
- Albany Medical Center, Albany, New York, United States

IPD SHARING:
Plan to Share IPD: No